CLINICAL TRIAL: NCT04551521
Title: Continuous ReAssessment With Flexible ExTension in Rare Malignancies - CRAFT: The NCT-PMO-1602 Phase II Trial
Brief Title: CRAFT: The NCT-PMO-1602 Phase II Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: German Cancer Research Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCT-PMO-1602
Record Dates: First submitted 2020-07-24; First posted 2020-09-16 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-05

CONDITIONS: Metastatic or Locally Advanced Malignancies
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Vemurafenib; cobimetinib; atezolizumab; Trastuzumab; pertuzumab; alectinib; ipatasertib; inavolisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- BRAF V600E/K (Experimental)
  Interventions: Drug: Vemurafenib; Drug: Cobimetinib; Drug: Atezolizumab
- ERBB2 (Experimental)
  Interventions: Drug: Trastuzumab; Drug: Pertuzumab; Drug: Atezolizumab
- ALK (Experimental)
  Interventions: Drug: Alectinib
- AKT/PTEN (Experimental): Recruitment stopped
  Interventions: Drug: Ipatasertib; Drug: Atezolizumab
- PI3K (Experimental): Recruitment stopped
  Interventions: Drug: Inavolisib
- MAPK (Experimental)
  Interventions: Drug: Cobimetinib; Drug: Atezolizumab
- Immune evasion (Experimental)
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Vemurafenib — 960 mg twice daily during run-in Phase, followed by 720 mg twice daily
  Arms: BRAF V600E/K
Drug: Cobimetinib — 60 mg once daily
  Arms: BRAF V600E/K; MAPK
Drug: Atezolizumab — 840 mg every 2 weeks
  Arms: BRAF V600E/K; MAPK
Drug: Trastuzumab — 8 mg per kilogram of body weight as a loading dose, followed by 6 mg per kilogram every 3 weeks
  Arms: ERBB2
Drug: Pertuzumab — 840 mg as a loading dose, followed by 420 mg intravenously every 3 weeks
  Arms: ERBB2
Drug: Alectinib — 600 mg twice daily
  Arms: ALK
Drug: Ipatasertib — 400 mg once daily
  Arms: AKT/PTEN
Drug: Atezolizumab — 1200 mg every 3 weeks
  Arms: ERBB2
Drug: Atezolizumab — 1200 mg in the first cycle, followed by 840 mg every 3 weeks
  Arms: AKT/PTEN
Drug: Atezolizumab — 1,200 mg every 3 weeks
  Arms: Immune evasion
Drug: Inavolisib — 9 mg once daily
  Arms: PI3K

SUMMARY:
Whole-genome and transcriptome sequencing of patients with advanced solid tumors enrolled in the NCT/DKTK MASTER (Molecularly Aided Stratification for Tumor Eradication Research) program revealed genetic alterations in a substantial proportion of patients including (i) alterations that lead to aberrant activation of BRAF, ERBB2, ALK, and the PI3K-AKT and MAPK pathways and (ii) changes that predict sensitivity to immune checkpoint inhibition, such as high tumor mutational burden and specific alterations of the PD-L1 locus.

Within this seven-arm basket phase II clinical trial, we aim to investigate the efficacy of targeted-therapy plus immune checkpoint inhibition in patients with advanced tumors exhibiting one of the following genetic alterations detected within the NCT/DKTK MASTER study: (i) BRAF V600E/K, (ii) ERBB2 amplification and/or overexpression or activating ERBB2 mutation, (iii) ALK rearrangement or activating ALK mutation, (iv) activating mutations or amplification of AKT, loss of PTEN, (v) activating PIK3CA mutations, (vi) abberations predicting increased RAF-MEK-ERK pathway activity; (vii) patients with high tumor mutational burden and/or specific alteration predicting sensitivity to PD-1/PD-L1 inhibition are eligible within this study for immune checkpoint inhibition. Recruitment of adequate patient numbers into these well-defined molecular subgroups is achieved in a multicenter approach including NCT Heidelberg and NCT Dresden as well as DKTK partner sites. Eligible patients will be identified by in-depth molecular characterization of tumors within the NCT/DKTK MASTER program. All study arms are based on similar biometrical assumptions, and sample size as well as power calculations are based on Simon's optimal two-stage design for each study arm separately. The overall aim is to reduce the cumulative hazard of progression-free survival observed within the study (PFS2) compared to the cumulative hazard of the progression-free time before inclusion into the study (PFS1) using a paired log-rank test. The sample size of the entire trial varies according to the performance of the individual study arms, ranging between 98 and 175 patients.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Ability of patient to understand and comply with the protocol for the duration of the study, including treatment and scheduled visits and examinations
* Diagnosis of a metastatic or locally advanced malignancy
* Progressive disease
* At least one measurable lesion that can be accurately assessed at baseline by computed tomography or magnetic resonance imaging and is suitable for repeated assessment
* Prior administration of at least one standard chemotherapy for primary and/or relapsed malignancy according to current guidelines. Patients must have received standard therapy or have no standard therapy available. Or, in the opinion of investigator have been considered ineligible for a particular form of standard therapy on medical reasons.
* ECOG Performance Status ≤2
* Age ≥18 years, no upper age limit
* Postmenopausal or evidence of non-childbearing status.
* Female patients of childbearing potential and male patients with partners of childbearing potential who are sexually active must agree to the use of two highly effective forms of contraception. These should be started immediately after signing the informed consent form and continued throughout the period of study treatment plus at least seven months for both sexes after taking the last dose of study drug.
* Availability of complete information about the last medical treatment given before study participation, i.e. remission status before start of treatment, dosage and timing of drugs applicated, remission status and date of progression after treatment (in order to calculate PFS 1)
* For patients included on the basis of molecular testing other than NCT/DKTK MASTER and for patients with an analysis in NCT/DKTK MASTER performed more than 3 months (date of tissue sampling) before planned study inclusion, a new tumor biopsy before start of study treatment is mandatory. However, patients may be included in the trial with archival tissue not older than 3 months on the basis of a case by case discussion with the PI.

Arm-specific Inclusion Criteria as determined by Whole Genome Sequencing and RNA Sequencing in NCT/DKTK MASTER or identification by gene panel performed in a certified lab Eligibility for the trial and the respective trial arms will be evaluated and determined exclusively by the NCT/DKTK molecular tumor board on the basis of results from NCT/DKTK MASTER (for all arms) or of results from other molecular studies, e.g. gene panel testing, performed in a certified laboratory (for arms 1-6). Trial participation is only possible with a report of the NCT/DKTK MASTER MTB confirming trial eligibility.

* Arm 1 (BRAF V600E/K): BRAF V600E/K mutation
* Arm 2 (ERBB2): ERBB2 amplification/overexpression, activating ERBB2 mutation
* Arm 3 (ALK): ALK rearrangement or activating ALK mutations including alternative transcription initiation (ALK-ATI) or RET-fusions
* Arm 4 (AKT/PTEN): Activating AKT1/2/3 mutations or amplifications; PTEN loss
* Arm 5: (PI3K): Activating PIK3CA mutations
* Arm 6 (MAPK): Aberrations other than BRAF V600E/K predicting increased RAF-MEK- ERK pathway activity
* Arm 7 (Immune evasion): High tumor mutational burden and/or specific alterations predicting sensitivity to PD1/PDL1 inhibition (e.g. DNA mismatch repair deficiency or PDL1 amplification and/or overexpression), ineligibility for the six specific arms

Exclusion Criteria (general):

* Other malignancy except for study indication within the last 5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), Stage 1, grade 1 endometrial carcinoma, or other malignancies curatively treated with no evidence of disease for ≥5 years
* Concurrent or previous treatment within 30 days prior to C1D1 in another interventional clinical trial with an investigational anticancer therapy
* Persistent toxicity (≥Grade 2 according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0) caused by previous cancer therapy, excluding alopecia
* Clinical signs of active infection (>Grade 2 according to CTCAE version 5.0)
* History of human immunodeficiency virus (HIV) infection and immunocompromised patients
* Active Hepatitis A virus infection
* Active hepatitis B virus (HBV) infection, defined as having a positive hepatitis B surface antigen (HBsAg) test at baseline patients with a past or resolved HBV infection, defined as having a negative HBsAg test and a positive total hepatitis B core antibody (HBcAb) test at baseline , are eligible for the study if active HBV infection is ruled out on the basis of HBV DNA viral load per local guidelines
* Active hepatitis C virus (HCV) infection, defined as having a positive HCV antibody test at baseline confirmed by a polymerase chain reaction (PCR) positive for HCV RNA
* Dementia or significant impairment of cognitive state
* Epilepsy requiring pharmacologic treatment
* Pregnancy or breastfeeding
* Inability to take oral medication orgastrointestinal disorders likely to interfere with absorption of the study medication (except Arm 2 and Arm 7)
* Major surgery within four weeks of starting study treatment
* Systemic chemotherapy or radiotherapy within two weeks prior to start of study treatment or a longer period depending on the characteristics of the agents used (at least five-half lives)
* Heart failure New York Heart Association (NYHA) II/III/IV
* Severe obstructive or restrictive ventilation disorder
* Prior allogeneic bone marrow transplantation or solid organ transplant.
* Administration of a live, attenuated vaccine within 4 weeks before initiation of study treatment or anticipation that such a live attenuated vaccine will be required during the study
* Patients with clinical suspicion of active tuberculosis
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug
* Is taking or requiring the continued use of any of the prohibited concomitant medications listed in the trial protocol
* Any concurrent antineoplastic therapy.
* Known suspected active alcohol or drug abuse
* Hematological malignancies and primary brain tumors. Patients with known progressive brain metastases determined by serial imaging or declining neurologic function in the opinion of the treating physician are not eligible. Patients with symptomatic uncontrolled brain metastases and patients with symptomatic uncontrolled spinal cord compression are not eligible. Patients with previously treated brain metastases are eligible, provided that the patient has not experienced a seizure or had a clinically significant change in neurological status within the three months prior to enrollment. All patients with previously treated brain metastases must be clinically stable for at least 1 month after completion of treatment and off steroid treatment for one month, both prior to study enrolment. Patients with asymptomatic untreated CNS disease may be enrolled, provided all of the following criteria are met:

  * Evaluable or measurable disease outside the CNS
  * No metastases to brain stem, midbrain, pons, medulla, cerebellum, or within 10 mm of the optic apparatus (optic nerves and chiasm)
  * No history of intracranial hemorrhage or spinal cord haemorrhage
  * No ongoing requirement for dexamethasone for CNS disease; patients on a stable dose of anticonvulsants are permitted
* Immune disease as specified below (relevant for all patients at Baseline except arm 3 and 5 (Alectinib, Inavolisib))

  * History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis; autoimmune-related hypothyroidism (patients on a stable dose of thyroid replacement hormone are eligible for this study) and type I diabetes mellitus (patients on a stable dose of insulin regimen are eligible for this study).
  * History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or active pneumonitis; history of radiation pneumonitis in the radiation field (fibrosis) is permitted.
  * Psoriatic arthritis (however, patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only are permitted provided that they meet the following conditions:
  * Rash must cover less than 10% of body surface area (BSA)
  * Disease is well controlled at baseline and only requiring low potency topical steroids
  * No acute exacerbations of underlying condition within the previous 12 months (not requiring PUVA [psoralen plus ultraviolet A radiation], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, high potency or oral steroids]).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Disease Control Rate | Day 110 (+/- 5 days)
  Primary endpoint of the study is to DCR according to RECIST v1.1 including complete response (CR), partial response (PR) and stable disease (SD).

SECONDARY OUTCOMES:
Progression-free survival | 24 months (median)
  Paired Progression-free Survival 2 (PFS2) and Progression-free Survival 1 (PFS1)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Schlenk, Prof. Dr., Study Director — NCT Studienzentrale
Locations (9):
- Germany (9):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Nationales Centrum für Tumorerkrankungen (NCT), Dresden
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Nationales Centrum für Tumorerkrankungen (NCT), Heidelberg
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Universitätsmedizin der Johannes Gutenberg- Universität Mainz, Mainz
  - Klinikum Rechts der Isar der TU München, München
  - Universitätsklinikum Tübingen, Medizinische Klinik I, Tübingen
  - Universitätsklinikum Würzburg, Interdisziplinäres Studienzentrum mit ECTU, Würzburg

REFERENCES:
- [Derived] Heilig CE, Horak P, Kreutzfeldt S, Teleanu V, Mock A, Renner M, Bhatti IA, Hutter B, Hullein J, Frohlich M, Uhrig S, Susse H, Heiligenthal L, Ochsenreither S, Illert AL, Vogel A, Desuki A, Heinemann V, Heidegger S, Bitzer M, Scheytt M, Brors B, Hubschmann D, Baretton G, Stenzinger A, Steindorf K, Benner A, Jager D, Heining C, Glimm H, Frohling S, Schlenk RF. Rationale and design of the CRAFT (Continuous ReAssessment with Flexible ExTension in Rare Malignancies) multicenter phase II trial. ESMO Open. 2021 Dec;6(6):100310. doi: 10.1016/j.esmoop.2021.100310. Epub 2021 Nov 20. PMID 34808524